CLINICAL TRIAL: NCT02071446
Title: Local Field Potentials Recorded From Deep Brain Stimulating Electrodes Implanted for the Treatment of Parkinson's Disease, Essential Tremor or Dystonia
Brief Title: Local Fields Potentials Recorded From Deep Brain Stimulating Electrodes
Acronym: LFP DBS
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Houston (Other); U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 13-3197
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Parkinson's Disease; Essential Tremor; Dystonia
Keywords: Deep Brain Stimulation; Local Field Potential; Subthalamic Nucleus
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Deep Brain Stimulation (DBS) is an FDA approved, and widely used method for treating the motor symptoms of Parkinson's Disease (PD), Essential Tremor (ET) and Dystonia. Over 100,000 patients worldwide have now been implanted with DBS devices. The DBS target regions in the brain are the Subthalamic nucleus (STN), the Internal Segment of Globus Pallidus (GPi), or the Ventral Intermediate Nucleus of the Thalamus (VIM). In order to place the DBS electrode in the target location, a combination of two 3D imaging techniques; 3D MRI and CT, are used. Data are also collected from individual nerve cells to help find the best location for the DBS electrode in each patient. This electrode recording takes place during the standard surgical implantation of the DBS electrode, and is part of the standard clinical technique. The investigators plan to collect additional data from populations of neurons during the DBS surgery in an effort to further improve the placement of the DBS electrode. These "Local Field Potentials", LFPs, represent the activity of the collection of neurons surrounding the tip of the electrode, and will be measured during surgery along the path used for the placement of the DBS electrode. The goal of this project is to determine whether this additional data from surrounding neurons will help with optimal placement of the DBS electrode.

ELIGIBILITY:
Inclusion Criteria:

* Subjects included in this study will be those who are planning to undergo DBS surgery because of their underlying idiopathic Parkinson's disease, Essential Tremor, or Dystonia--all FDA-approved indications for the implantation of DBS devices.

Exclusion Criteria:

* Subjects with the most advanced symptoms of PD (stage V in the Hoehn and Yahr rating scale).
* Subjects who are not planning to undergo DBS surgery.
* Subjects not candidates for DBS surgery based on clinical criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Movement disorder patients from primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Recording and evaluating LFPs from DBS electrodes | at baseline
  Recording and evaluating LFPs from DBS electrodes in patients with Parkinson's Disease, Essential Tremor or Dystonia

CONTACTS AND LOCATIONS:
Overall Officials: Aviva Abosch, MD, PhD., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States